CLINICAL TRIAL: NCT02293993
Title: Phase 1 Study of SGI-110 in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 343-14-001; JapicCTI-142711 (Other: Japic)
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort1 (Experimental): SGI-110 36mg/m2 will be administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
  Interventions: Drug: SGI-110
- Cohort2 (Experimental): SGI-110 60mg/m2 will be administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
  Interventions: Drug: SGI-110
- Cohort3 (Experimental): SGI-110 90mg/m2 will be administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
  Interventions: Drug: SGI-110
- Cohort4 (Experimental): SGI-110 60mg/m2 will be administered subcutaneously once daily for 10 days (Day 1 to Day 5 and Day 8 to Day 12 with dosing, Day 6 and 7 with non-dosing), followed by a 16-day non-dosing period (Day 13 to Day 28).
  Interventions: Drug: SGI-110

INTERVENTIONS:
Drug: SGI-110

SUMMARY:
To evaluate the tolerability and pharmacokinetics of SGI-110 when administered subcutaneously to Japanese patients with acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a diagnosis of AML (WHO classification 2008).

  * Patients, 20 years of age or older, who are unresponsive to standard chemotherapy or have relapsed following standard chemotherapy
  * Patients, 65 years of age or older, who are not eligible for standard intensive chemotherapy
* Patients with ECOG performance status (PS) of 0 to 2
* Patients with adequate organ function
* Women of child-bearing potential must not be pregnant or breast feeding (pregnancy test will be performed at Screening). Women of child bearing potential and all men with female partners of child bearing potential must practice two medically acceptable methods of birth control and must not become pregnant or father a child while receiving treatment with SGI-110 and for 3 months following last dosing.
* Patients who have undergone prior allogeneic hematopoietic stem cell transplantation must have no evidence of active graft-versus host disease (GVHD) and must be off immunosuppressive therapy by ≥2 weeks prior to IMP administration.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia accompanied by t(15;17)(q22;q12) or (PML/RARA) karyotype abnormalities (include other variant types of APL)
* Patients with multiple cancers (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for at least 3 years)
* Subjects with life-threatening illnesses other than AML or MDS, uncontrolled medical conditions or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, or put the study outcomes at risk.
* Patients with poorly controlled arrhythmias, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Patients with symptomatic central nervous system involvement.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junji Ikeda, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (3):
- Japan (3):
  - kinki Region, Kyoto
  - Kanto, Region
  - Kyusyu, Region

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial consisted of a screening period, dose limiting toxicity (DLT) evaluation period (Course 1), and withdrawal examination. Subjects who completed investigational medicinal product (IMP) administration and all observations during the DLT evaluation period, and who did not have any apparent progression of AML, were permitted to be added extended treatment period (Course 2) to continue treatment with IMP following the DLT evaluation period if they wished.
Groups:
- Cohort 1: SGI-110 36mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
- Cohort 2: SGI-110 60mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
- Cohort 3: SGI-110 60mg/m2 was administered subcutaneously once daily for 10 days in total (Day 1 to Day 5 and Day 8 to Day 12 with dosing, Day 6 and 7 with non-dosing), followed by a 16-day non-dosing period (Day 13 to Day 28).
- Cohort 4: SGI-110 90mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
Period: Course 1 (DLT Evaluation Period)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 4 | 6 | 7 | 4
Completed | 3 | 6 | 7 | 3
Not Completed | 1 | 0 | 0 | 1
Not completed — Clear progression of the primary disease including relapses | 1 | 0 | 0 | 1
Period: Course ≥2 (Extended Treatment Period)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 2 | 5 | 6 | 3
Completed | 0 | 0 | 1 | 2
Not Completed | 2 | 5 | 5 | 1
Not completed — Physician Decision | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Clear progression of the primary disease including relapses | 2 | 2 | 3 | 1
Not completed — Delay in commencement of the next course by more than 4 weeks | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included subjects who had received at least one dose of the IMP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 4 | 6 | 7 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 3 | 6 | 7 | 4 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 1 | 9
  Male | 2 | 5 | 2 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 4 | 6 | 7 | 4 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 6 | 7 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: DLT was defined as any of the following adverse events (AEs) occurring during Course 1 for which there was a reasonable probability or possibility of a causal relationship with the IMP. The severity of AEs was graded in accordance with Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  * Nonhematologic toxicity of Grade ≥3, except for (i) nausea, vomiting, or diarrhea of Grade 3 that is controllable by optimal therapy, and (ii) Grade 3 laboratory findings other than serum creatinine, bilirubin, aspartate aminotransferase, or alanine aminotransferase.
  * Grade 4 thrombocytopenia that was not present at trial entry and that is not resolved within 7 days
  * Grade 4 neutropenia that was not present at trial entry and that is not resolved within 7 days
  * Febrile neutropenia (defined as a neutrophil count of <500/μL accompanied by a fever of ≥38°C)
  * Any AE that results in a delay of >4 weeks in starting the next treatment course
Time Frame: 28 days (Day 1 to Day 29)
Population: DLT analysis population included subjects in whom tolerability had been assessed in Cohorts 1 to 4 (subjects who had received all doses and completed all assessments scheduled for the DLT evaluation period).
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 6 | 6 | 3
participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SGI-110 and Its Active Metabolite Decitabine Following Single and Multiple Administration of SGI-110
Time Frame: Pre-dose, 15min, 30min, 60min, 90min, 2h, 3h, 4h, 6h, 8h, 24h after dosing (Cohorts 1, 2, and 4: Day 1 and Day 5, Cohort 3: Day 1 and Day 12)
Population: Analysis population included subjects whose plasma drug concentrations had been measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1 (Day 1); Cohort 1 (Day 5): SGI-110 36mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
- Cohort 2 (Day 1); Cohort 2 (Day 5): SGI-110 60mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
- Cohort 3 (Day 1); Cohort 3 (Day 12): SGI-110 60mg/m2 was administered subcutaneously once daily for 10 days in total (Day 1 to Day 5 and Day 8 to Day 12 with dosing, Day 6 and 7 with non-dosing), followed by a 16-day non-dosing period (Day 13 to Day 28).
- Cohort 4 (Day 1); Cohort 4 (Day 5): SGI-110 90mg/m2 was administered subcutaneously once daily for 5 consecutive days (Day 1 to Day 5), followed by a 23-day non-dosing period (Day 6 to Day 28).
Arm/Group | Cohort 1 (Day 1) | Cohort 2 (Day 1) | Cohort 3 (Day 1) | Cohort 4 (Day 1) | Cohort 1 (Day 5) | Cohort 2 (Day 5) | Cohort 3 (Day 12) | Cohort 4 (Day 5)
Number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 7 | 4
ng/mL
  SGI-110: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  SGI-110 | 96.8 (37.3) | 182 (59.7) | 140 (33.1) | 359 (220) | 142 (97.4) | 200 (42.4) | 155 (58.5) | 328 (208)
  decitabine: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  decitabine | 28.6 (13.8) | 54.1 (14.7) | 31.8 (4.08) | 109 (50.3) | 38.2 (34.1) | 67.2 (13.5) | 44.5 (15.3) | 95.7 (37.2)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of SGI-110 and Its Active Metabolite Decitabine Following Single and Multiple Administration of SGI-110
Time Frame: as for outcome 2
Population: Analysis population included subjects whose plasma drug concentrations had been measured.
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 (Day 1) | Cohort 2 (Day 1) | Cohort 3 (Day 1) | Cohort 4 (Day 1) | Cohort 1 (Day 5) | Cohort 2 (Day 5) | Cohort 3 (Day 12) | Cohort 4 (Day 5)
Number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 7 | 4
h
  SGI-110: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  SGI-110 | 1.49 [0.48 to 1.50] | 0.98 [0.23 to 1.45] | 1.48 [0.53 to 1.98] | 1.51 [0.50 to 2.85] | 0.99 [0.48 to 1.50] | 0.97 [0.52 to 2.00] | 1.42 [0.97 to 1.48] | 1.27 [0.48 to 3.00]
  decitabine: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  decitabine | 2.04 [0.48 to 3.02] | 1.27 [0.52 to 1.50] | 1.93 [1.03 to 2.00] | 1.51 [1.02 to 2.85] | 1.49 [0.48 to 2.00] | 1.47 [0.92 to 2.00] | 1.43 [0.97 to 2.02] | 1.53 [1.00 to 3.00]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC24h) of SGI-110 and Its Active Metabolite Decitabine Following Single and Multiple Administration of SGI-110
Time Frame: as for outcome 2
Population: Analysis population included subjects whose plasma drug concentrations had been measured.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Cohort 1 (Day 1) | Cohort 2 (Day 1) | Cohort 3 (Day 1) | Cohort 4 (Day 1) | Cohort 1 (Day 5) | Cohort 2 (Day 5) | Cohort 3 (Day 12) | Cohort 4 (Day 5)
Number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 7 | 4
ng·h/mL
  SGI-110: number analyzed (Participants) | 4 | 6 | 7 | 3 | 4 | 5 | 6 | 4
  SGI-110 | 207 (36.1) | 398 (75.7) | 332 (61.5) | 710 (119) | 206 (11.7) | 410 (57.9) | 311 (87.2) | 581 (124)
  decitabine: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  decitabine | 70.0 (13.4) | 151 (42.7) | 95.7 (11.7) | 248 (39.9) | 67.0 (18.6) | 150 (34.1) | 101 (10.7) | 240 (41.6)

5. Secondary Outcome: Terminal-phase Elimination Half-life (T1/2,z) of SGI-110 and Its Active Metabolite Decitabine Following Single and Multiple Administration of SGI-110
Time Frame: as for outcome 2
Population: Analysis population included subjects whose plasma drug concentrations had been measured.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 (Day 1) | Cohort 2 (Day 1) | Cohort 3 (Day 1) | Cohort 4 (Day 1) | Cohort 1 (Day 5) | Cohort 2 (Day 5) | Cohort 3 (Day 12) | Cohort 4 (Day 5)
Number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 7 | 4
h
  SGI-110: number analyzed (Participants) | 4 | 6 | 7 | 3 | 4 | 5 | 6 | 4
  SGI-110 | 0.698 (0.393) | 0.833 (0.493) | 0.740 (0.212) | 0.656 (0.155) | 0.599 (0.332) | 0.503 (0.144) | 0.685 (0.341) | 0.623 (0.153)
  decitabine: number analyzed (Participants) | 4 | 6 | 7 | 4 | 4 | 6 | 6 | 4
  decitabine | 1.04 (0.467) | 1.12 (0.564) | 1.09 (0.148) | 0.891 (0.0990) | 0.905 (0.385) | 0.821 (0.231) | 1.14 (0.486) | 0.875 (0.107)

ADVERSE EVENTS:
Time Frame: From the start of IMP administration up to 5 days after withdrawal
Description: A treatment-emergent adverse event (TEAE) was defined as an AE occurring after the start of IMP administration.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/6 | 4/7 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=4)
Lung infection (Infections and infestations) | 0 | 2 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=4)
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Trichophytosis (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3 | 0
Sleep disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Internal haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Senile pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Genital erosion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Genital ulceration (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 1
Injection site induration (General disorders) | 0 | 3 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 1
Injection site erythema (General disorders) | 0 | 2 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Injection site vesicles (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 3 | 0
Lymphocyte count decreased (Investigations) | 1 | 5 | 6 | 3
Platelet count decreased (Investigations) | 2 | 1 | 6 | 3
White blood cell count decreased (Investigations) | 2 | 1 | 4 | 2
Neutrophil count decreased (Investigations) | 2 | 1 | 2 | 1
Weight decreased (Investigations) | 0 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 1
Reticulocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1
Antithrombin III decreased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT02293993/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT02293993/SAP_001.pdf